CLINICAL TRIAL: NCT07204496
Title: A Clinical Study on the Safety, Tolerance, and Preliminary Efficacy of γδ-T Cell Injection in the Treatment of Advanced Bladder Cancer
Acronym: γδ-T-BLADDER
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Wei Li, M.D., Shanghai 10th People's Hospital
Other Study IDs: SHSY-IEC-6.0/24K176/P02
Record Dates: First submitted 2025-09-04; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Advanced Bladder Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Advanced Bladder Cancer
  Interventions: Biological: Ex Vivo Expanded γδ T Cell Infusion

INTERVENTIONS:
Biological: Ex Vivo Expanded γδ T Cell Infusion — This study involves the use of γδ T cell infusion, a non-genetically modified adoptive cellular immunotherapy. The intervention utilizes autologous γδ T cells isolated from peripheral blood and expanded ex vivo using specific activators such as zoledronate and cytokines, without genetic engineering. Its mechanism of action relies on the inherent MHC-unrestricted tumor recognition capability of γδ T cells, activating both the NKG2D-NKG2DL axis and BTN3A1-CD277 pathway for dual antitumor activity. The manufacturing process follows GMP-compliant closed-system conditions, with final product release criteria requiring ≥80% purity for CD3+γδ TCR+ cells, along with sterility testing, endotoxin detection, and cytotoxicity assays. This approach fundamentally differs from genetically modified αβ T cell-based therapies like CAR-T or TCR-T, as well as non-specific immunotherapies such as CIK/DC-CIK, and demonstrates superior ex vivo expansion and tumor-targeting capabilities compared to TIL therap

SUMMARY:
We plan to enroll 20-29 patients with advanced bladder cancer to undergo T-cell therapy. Each treatment cycle consists of three T-cell infusions, with two cycles planned per patient. Each cycle will include imaging studies, laboratory tests, and vital sign monitoring to evaluate quality of life and treatment efficacy. Through real-world clinical data, we aim to scientifically determine whether this novel T-cell therapy can significantly alter the pathological progression of tumors and improve patient outcomes. Ultimately, we seek to benefit a broader patient population by achieving long-term tumor-bearing or tumor-free survival, transforming cancer management into a chronic disease model and improving patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

The subject voluntarily participates in this study, signs the informed consent form, demonstrates good compliance, and agrees to follow-up.

Aged 18-75 years, regardless of gender.

Diagnosed with primary bladder cancer confirmed by histopathology or clinical diagnostic criteria, clinically assessed as unresectable, and having failed at least two prior lines of standard therapy.

Adequate organ function:

1. Hematologic system (no transfusion or hematopoietic growth factor therapy within 14 days prior to enrollment):

   Absolute neutrophil count (ANC) ≥1.5×10⁹/L

   Platelets (PLT) ≥60×10⁹/L

   Hemoglobin (Hb) ≥90 g/L
2. Liver function:

   Total bilirubin (TBIL) ≤1.5×ULN

   Alanine aminotransferase (ALT) ≤3×ULN

   Aspartate aminotransferase (AST) ≤3×ULN

   Albumin ≥2.8 g/dL
3. Coagulation function:

   Activated partial thromboplastin time (APTT) ≤1.5×ULN

   International normalized ratio (INR) or prothrombin time (PT) within normal range
4. Renal function:

   Serum creatinine ≤1.5×ULN, or

   Creatinine clearance (Ccr) ≥50 mL/min (calculated using Cockcroft-Gault formula; applies only if creatinine >1.5×ULN)
5. Thyroid function:

   Thyroid-stimulating hormone (TSH) ≤1×ULN

   Free triiodothyronine (FT3) ≤1×ULN

   Free thyroxine (FT4) ≤1×ULN
6. Cardiovascular function:

Left ventricular ejection fraction (LVEF) ≥50% by echocardiography

AJCC Bladder Cancer Stage III or IV.

Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.

At least one measurable lesion (according to mRECIST criteria).

Expected survival time ≥6 months.

Male subjects with partners of childbearing potential must use reliable and effective contraception from signing the informed consent form until 180 days after the last dose of the study drug. Male subjects with pregnant partners must use condoms and require no additional contraception methods.

Exclusion Criteria:

Prior treatments within 28 days before the first dose:

1. Chemotherapy, radiotherapy, biologic therapy, immunotherapy, targeted therapy, local therapy, or traditional Chinese medicine with明确抗肿瘤适应症 (clear antitumor indications).
2. Major surgical procedures or failure to recover from side effects of such surgeries (excluding minor procedures, e.g., appendectomy, tumor biopsy).
3. Participation in other interventional drug clinical trials (excluding observational studies or survival follow-up).

Failure to recover from prior antitumor therapy-related toxicities (except alopecia) (i.e., toxicity still > Grade 1 or not returned to baseline).

Concurrent or history of other malignancies, except:

Curative basal cell or squamous cell skin cancer

Carcinoma in situ of the cervix

Papillary thyroid carcinoma

Ductal carcinoma in situ of the breast

Other malignancies with disease-free survival >5 years

Uncontrolled diabetes despite optimal supportive care.

Presence of gastrointestinal bleeding, refractory ascites, hepatic encephalopathy, or hepatorenal syndrome.

History or presence of autoimmune diseases (e.g., rheumatoid arthritis).

Neurological diseases, diffuse leptomeningeal disease, or comorbid neurodegenerative disorders.

History or planned stem cell or organ transplantation during the study.

Any of the following within 6 months before the first dose:

1. Cerebrovascular accident, transient ischemic attack, symptomatic pulmonary embolism, or other clinically significant thromboembolic events.
2. Unstable angina, myocardial infarction, or symptomatic chronic heart failure.
3. Ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes).
4. Coronary/peripheral artery bypass grafting.
5. Current or history of congestive heart failure (NYHA Class II-IV).
6. Uncontrolled hypertension despite medication (systolic BP ≥160 mmHg and/or diastolic BP ≥100 mmHg).

Active infections, including:

1. Clinically uncontrolled active infections within 7 days before the first dose (e.g., acute pneumonia, unexplained persistent fever).
2. Hepatitis B (HBsAg-positive and HBV-DNA >1000 IU/mL; HBV carriers must receive antiviral therapy per local guidelines and commit to ongoing treatment during the study).
3. Hepatitis C (HCV antibody-positive).
4. HIV or Treponema pallidum (TP) infection.

Requirement for systemic corticosteroids (>10 mg/day prednisone or equivalent) or other immunosuppressants.

Pregnancy or lactation.

Any uncontrolled concurrent condition (including psychiatric disorders or substance abuse) deemed by the investigator to compromise subject cooperation or trial participation, or any other reason making the subject unsuitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from adult patients (aged 18-75 years) with histologically confirmed, unresectable advanced bladder cancer (AJCC Stage III or IV) who have failed at least two prior lines of standard therapy. The population will include individuals with adequate organ function (hematologic, hepatic, renal, cardiac, and coagulation parameters per predefined criteria) and an ECOG performance status of 0-1. Key exclusions comprise active autoimmune diseases, uncontrolled infections, concurrent malignancies, organ transplant recipients, and significant cardiovascular/neurological comorbidities. This trial specifically targets a population eligible for investigational cellular immunotherapy, focusing on those with progressive disease despite conventional treatments.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-09-26 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From the time of randomization (or initiation of treatment) until the occurrence of objective tumor progression or death from any cause, whichever occurs first.
Progression-Free Survival (PFS) | From enrollment to the end of treatment at 30 days

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol